CLINICAL TRIAL: NCT01661192
Title: Open Label Study (Extension 001)to Evaluate Long Term Treatment Effect of the Safety, Tolerability and Efficacy of Intervenous ALPHA-1 ANTITRYSIN (AAT)Glasia™ in Type 1 Diabetes Mellitus (Extension to KAMADA AAt 008, PHASE I/II Study)
Brief Title: Long Term Treatment Effect of the Safety, Tolerability and Efficacy of AAT in Type 1 Diabetes
Acronym: AAT Extension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 006971ctil
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Type 1 Diabetes; Beta Cell Preservation
Keywords: Type 1 Diabetes; newly diagnosed; Beta cell preservation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — alpha 1-antitrypsin-leukocyte elastase complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AAT( Alpha 1 Antitrypsin) (Experimental): Subjects who maintained peak stimulated C-peptide secretion ≥ 0.2nmol/L will continue treatment with AAT according to the dosage group they were allocated to at the previous study(40mg/kg or 60mg/kg or 80mg/kg), intravenously, once a week for 6 consecutive weeks, at 24-week intervals for a duration of ~54 weeks.
  Interventions: Drug: AAT( Alpha 1 Antitrypsin)
- Follow up group (No Intervention): Subjects who have not maintained peak stimulated C-peptide secretion ≥ 0.2nmol/L or subjects with peak stimulated C -peptide secretion ≥ 0.2nmol/L who are reluctant to receive additional study drug, will be followed up only with no administration of investigational product

INTERVENTIONS:
Drug: AAT( Alpha 1 Antitrypsin)
  Arms: AAT( Alpha 1 Antitrypsin)

SUMMARY:
At a previous study the investigators have assessed the safety and efficacy of treatment with AAT(Alpha 1 Antitrypsin)in newly diagnosed type 1 diabetes subjects aiming at beta cells preservation .

Since treatment with AAT is expected to be a chronic treatment; stopping treatment will probably result in eventual loss of the preserved beta-cell function. Indeed, other investigational drugs aiming at beta cells preservation have shown that patients who were initially treated and maintained their initial beta-cell function, required continuation of treatment or they lost the beta-cell function.

Therefore, in this extension study, patients who were previously treated with AAT and maintained clinically significant beta-cell function are offered a continuation of treatment, since they are likely to benefit from use of the medication.

The proposed study is aimed to assess the long term effect of AAT in subjects with type 1 diabetes mellitus: safety and tolerability of treatment, and effect on beta-cell function.

Subjects who have completed all visits of the 008 study will be offered to participate in the extension study.

The study will be consist off two main arms as following:

Arm 1: Subjects who maintained peak stimulated C-peptide secretion ≥ 0.2 nmol/L will continue treatment with AAT for up to 18 treatments according to the dosage group they were allocated to in the 008 study.

Arm 2:

Subjects who have not maintained peak stimulated C-peptide secretion ≥ 0.2nmol/L and subjects with peak stimulated C -peptide secretion ≥ 0.2 nmol/L who are reluctant to receive additional study drug.

Clinical follow up for all subjects in both arms will be for 3 years

ELIGIBILITY:
Inclusion Criteria:

* Subject (or parent/guardian) willing and able to sign an informed consent
* Ability to comply with all study requirements.
* A patient that participated in Study 008 and received all doses of study medication, per protocol.
* Evidence of clinically significant residual beta-cell function demonstrated by MMTT peak stimulated C-peptide concentrations ≥ 0.20 nmol/L (Arm 1 only).
* Age 10-25 (inclusive) years
* If a female is of childbearing potential, the subject is not pregnant or lactating, and will use oral hormonal contraception or other equally effective contraceptive methods throughout the study.

Exclusion Criteria:

* IgA (immunoglobulin A ) deficient subjects.
* Individuals with a history of severe immediate hypersensitivity reactions, including anaphylaxis, to plasma products.
* History of life threatening allergy, anaphylactic reaction, or systemic response to human plasma derived products.
* The subject is receiving immunosuppressive or immunomodulating agents or cytotoxic therapy or any medication that in the opinion of the Investigator might interfere with the study.
* Clinically significant intercurrent illnesses, including (but not limited to): cardiac, hepatic, renal, neurological, hematological, neoplastic, immunological, skeletal or other) that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study. Patients with well-controlled, chronic diseases could be possibly included after consultation with the treating physician.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AAT in terms of adverse events and serious adverse events | At month 36
  We will assess at each visit until final visit (month 36)the safety and tolerability of study drug in terms of adverse events and serious adverse events
Safety and tolerability of the AAT in terms of laboratory values | At month 36
  We will assess at each visit until final visit (month 36)the safety and tolerability of study drug in terms of laboratory values

SECONDARY OUTCOMES:
Beta cell function-AUC (Area Under the Curve) of stimulated C-Peptide from stimulated MMTT (mixed meal tolerance test) | at month 36
Percentage of patients that maintain stimulated peak C-peptide >=0.2 nmol/L | at month 36
Percentage of patients that achieve glycemic target of HbA1c <=7.5% | At month 36
Daily insulin dose adjusted to body weight | At month 36

CONTACTS AND LOCATIONS:
Overall Officials: Yael Lebenthal, MD, Principal Investigator — Rabin Medical Center; Mariana Rachmiel, MD, Principal Investigator — Assaf Haroffe Medical Center
Locations (2):
- Israel (2):
  - Schneider Children's Medical Center, Petah Tikva
  - Assaf Haroffeh Medical Center, Ẕerifin

REFERENCES:
- [Derived] Brener A, Lebenthal Y, Interator H, Horesh O, Leshem A, Weintrob N, Loewenthal N, Shalitin S, Rachmiel M. Long-term safety of alpha-1 antitrypsin therapy in children and adolescents with Type 1 diabetes. Immunotherapy. 2018 Sep;10(13):1137-1148. doi: 10.2217/imt-2018-0047. PMID 30236025